CLINICAL TRIAL: NCT06011408
Title: Remote Monitoring and Detecting of Tardive Dyskinesia for Improving Patient Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iRxReminder (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: #23-002; R43MH114763 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Intervention Model Description: Open-label, observational study with two groups taking antipsychotic with or without Tardive Dyskinesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taking antipsychotic medication with Tardive Dyskinesia (Other)
  Interventions: Other: TDtect
- Taking antipsychotic medication without Tardive Dyskinesia (Other)
  Interventions: Other: TDtect

INTERVENTIONS:
Other: TDtect — Collecting video data on abnormal movement

SUMMARY:
The study is being conducted to validate the feasibility of remote assessment of Tardive Dyskinesia.

DETAILED DESCRIPTION:
The study is being conducted to validate the feasibility of remote assessment of Tardive Dyskinesia. Participants will all be taking an antipsychotic medication and half will have a diagnosis of Tardive Dyskinesia and half will not. Participant responses to interview questions and elements of the Abnormal Involuntary Movement Scale will be collected on video. The videos will be rated by trained observers. Machine learning methods will be used to develop an algorithm to detect abnormal movements in individuals with a known Tardive Dyskinesia diagnosis. The trained rater results will be compared to the algorithm to determine the accuracy of the algorithm.

ELIGIBILITY:
Inclusion Criteria:

For the non-TD group:

1. Prescribed and taking an antipsychotic medication for 90-days or longer.
2. Tardive Dyskinesia symptoms if present are not from Parkinsons, Tourette's syndrome, Huntington disease.
3. Signed an informed consent.
4. Speaks English fluently.

Exclusion Criteria:

1. Suffered a moderate or severe head injury in the last year;
2. History of a learning disorder or developmental disability that would inhibit a patient from completing the TD protocol.
3. Severe visual impairment that is cannot be corrected by glasses or contacts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
AIMS Score | Baseline
  Abnormal Involuntary Scale Score

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Ranjan, M.D., Study Director — Charak Research Center; Owen Muir, M.D., Study Director — Fermata Health
Locations (2):
- United States (2):
  - Fermata Helath, Brooklyn, New York
  - Charak Research Center, Garfield Heights, Ohio

REFERENCES:
- See also: Related Info — http://www.irxreminder.com
- See also: Related Info — http://www.charakcenter.com
- See also: Related Info — http://www.fermata.health